CLINICAL TRIAL: NCT05072509
Title: Endoprothesis Long-term Behavior After Subrenal Abdominal Aortic Aneurysm
Brief Title: Assessment of the Endovascular Aortic Aneurysm Repair's (EVAR) Main Body Lateral Movement Impact on the Rate of Reintervention After AAA's Treatment
Acronym: COLONEA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Association Le Don du Souffle (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-598
Record Dates: First submitted 2021-08-16; First posted 2021-10-11 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2021-10

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: aortic; endovascular; aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The strength of movement which are applied on the EVAR are not only cranio-caudal but also lateral. The movement of the EVAR's body within the aneurysm could be an instability's criteria of the EVAR. The investigators would like to show that this lateral movement is a risk factor of reintervention they should follow and suggest a reinforced medical follow-up to avoid complications.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 18 years old
* All patients treated in the vascular surgery department of Besançon for an abdominal aortic aneurysm with an endoprothesis (symptomatic or asymptomatic)

Exclusion Criteria:

* Patient in emergency situation (ruptured abdominal aortic aneurysm)
* Life expectancy supposed to be inferior to 1 year
* Legal incapacity or limited capacity
* Pregnant female
* Patient unlikely to cooperate with the study
* Patient without health insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated in the vascular surgery department of Besançon for an abdominal aortic aneurysm with an endoprothesis (symptomatic or asymptomatic)
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Reintervention rate | through study completion, an average of 5 years
  For the the reintervention rate, all the intervention relative to a failure of the EVAR will be taken in account: as - Endoleak - Thrombosis - Conversion to open surgery - Infection - Secondary rupture
Lateral movement of the EVAR | through study completion, an average of 5 years
  The lateral movement is defined by a movement of more than 5 mm.

SECONDARY OUTCOMES:
EVAR's movements: other than lateral. | 1 month post-op, 6 months, 12 months, 2 years, 3 years, 4 years, 5 years.
  Other than lateral
Moving | 1 month post-op, 6 months, 12 months, 2 years, 3 years, 4 years, 5 years.
  EVAR's movement in relation to distal or proximal anchorage zones
Compliance | 1 month post-op, 6 months, 12 months, 2 years, 3 years, 4 years, 5 years.
  The number of CT scanner compared to the number recommended by the Haute Autorité de Santé (HAS)

CONTACTS AND LOCATIONS:
Locations (1):
- Vascular Surgery Department, Besançon, France